CLINICAL TRIAL: NCT01589419
Title: An Open-Label Phase 1b Study of the Safety and Tolerability of Veliparib in Combination With Capecitabine and Radiation in Subjects With Locally Advanced Rectal Cancer (LARC)
Brief Title: A Clinical Study Conducted in Multiple Centers Evaluating Escalating Doses of Veliparib in Combination With Capecitabine and Radiation in Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-950
Record Dates: First submitted 2012-04-30; First posted 2012-05-02 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2015-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: DLT; radiation; veliparib; locally advanced rectal cancer; ABT-888; capecitabine; MTD; PARP
MeSH Terms: interventions — veliparib; Capecitabine; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- veliparib and capecitabine and radiation (Experimental): Veliparib on days 1-7, capecitabine and radiation on days 1-5
  Interventions: Drug: veliparib; Drug: capecitabine; Radiation: radiation

INTERVENTIONS:
Drug: veliparib — see arm description
  Other Names: ABT-888
Drug: capecitabine — see arm description
  Other Names: Xeloda
Radiation: radiation — see arm description

SUMMARY:
An open-label, Phase 1b, dose escalation study evaluating the safety and tolerability of the PARP inhibitor Veliparib in combination with capecitabine and radiation in subjects with locally advanced rectal cancer (LARC).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 18 years of age
* All subjects must have newly diagnosed, histologically proven adenocarcinoma of the rectum
* All subjects must have an abdominal/pelvis computed tomography (CT ) scan or magnetic resonance imaging (MRI) confirming no evidence of distant metastases
* Distal border of tumor < 12 cm from anal verge
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 to 2
* No prior treatment for LARC however prior treatments for other cancers are acceptable as long as they are considered curative

Exclusion Criteria:

* Subject is an unsuitable candidate for TME surgery
* Subject has received anticancer therapy
* Subject has received prior radiation therapy
* Subject has had major surgery within 28 days prior to the first dose of study drug
* History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) and/or establish the recommended phase two dose (RPTD) | From first study drug dose and at each weekly treatment visit until dose-limiting toxicities (DLT) observed or completion of dosing period (anticipated to be approximately 5 weeks).

SECONDARY OUTCOMES:
Assess the safety (number of participants with adverse events and types of adverse events observed) | From screening and ongoing at each weekly treatment visit through dosing period (anticipated to be approximately 5 weeks), prior to surgery and at the final visit.
Assess the tolerability (number of participants with adverse events and types of adverse events observed) | From first study drug dose and ongoing at each weekly treatment visit, through completion of dosing period (anticipated to be approximately 5 weeks).
Assess the pharmacokinetic profile by area under the curve vs. dose of veliparib | Multiple measurements over time points (0, .5, 1, 2, 3, 4, 6 hours post dose) Day 1, Day 2 and at the pre-dose time point on Day 5 and week 2 visit.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Komarnitsky, MD, Study Director — AbbVie
Locations (6):
- United States (5):
  - Site Reference ID/Investigator# 99095, Scottsdale, Arizona
  - Site Reference ID/Investigator# 68044, Chicago, Illinois
  - Site Reference ID/Investigator# 112395, Goshen, Indiana
  - Site Reference ID/Investigator# 68045, Durham, North Carolina
  - Site Reference ID/Investigator# 68043, Madison, Wisconsin
- Site Reference ID/Investigator# 67882, East Melbourne, Australia

REFERENCES:
- [Result] Czito BG, Deming DA, Jameson GS, Mulcahy MF, Vaghefi H, Dudley MW, Holen KD, DeLuca A, Mittapalli RK, Munasinghe W, He L, Zalcberg JR, Ngan SY, Komarnitsky P, Michael M. Safety and tolerability of veliparib combined with capecitabine plus radiotherapy in patients with locally advanced rectal cancer: a phase 1b study. Lancet Gastroenterol Hepatol. 2017 Jun;2(6):418-426. doi: 10.1016/S2468-1253(17)30012-2. Epub 2017 Mar 27. PMID 28497757